CLINICAL TRIAL: NCT00886665
Title: The Evaluation of Safety and Efficacy of JWHGWT on Diabetic Neuropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Chia-I Tsai, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: grb03484777
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-04

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Nerve Conduction Studies; Clinical Trial
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- JWHGWT (Experimental)
  Interventions: Drug: JWHGWT

INTERVENTIONS:
Drug: placebo — placebo, 4 g, powder, oral, 3 times a day
  Arms: Placebo
Drug: JWHGWT — JWHGWT, 4 g, powder, oral, 3 times a day
  Arms: JWHGWT

SUMMARY:
In order to provide a alternative treatment for relieving the pain and numbness of Diabetes Mellitus patients,Traditional Chinese Medicine powder was tested by subjective questionnaire and objective nerve conduction velocity study. Liver and kidney functions were tested to provided safety profiles.

DETAILED DESCRIPTION:
120 participants with diabetic neuropathy were screened in endocrine and metabolism clinics of Taichung Veterans General Hospital and Chinese Medical University Hospital . Subjects were randomly distributed into a double-blind, 12 weeks, placebo-controlled procedure. Subjects were measured by MNSI, SF-BPI, SF-36, SF -MCQ, NCV, AC sugar, HbA1c, lipid profiles, liver and kidney functions.

Safety evaluations including GPT and creatinine revealed no deterioration after treatment. Several domains in MNSI, SF-BPI, SF-36, SF -MPQ questionnaires revealed significant improvements. F-wave in peroneal, tibial nerves and distal latency in tibial nerve in objective nerve conduction studies revealed significant improvements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of DM
* Must have the symptoms of pain or numbness

Exclusion Criteria:

* Patient with pregnancy (or child bearing potential),or in lactation
* Patient currently taking concomitant TCM medications.
* Patient with Drug or alcohol addiction
* Patient with medical history of myocardial infarction, cerebro-vascular disease, major trauma, operation 6 months prior to enrollment
* Patient with liver dysfunction (SGOT or SGPT>2x ULN)
* Patient with renal insufficiency (serum creatinine>1.3mg/dL)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Short-form (sf)- McGill pain questionnaire (SF-MPQ) | 0, 4, 8,12 weeks

SECONDARY OUTCOMES:
Nerve conduction study | 0,12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chia-I Tsai, master, Principal Investigator — Taichung Veterans General Hospital
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung, Taichung / Taichung
  - Taichung Veterans General Hospital, Taichung, Taichung

REFERENCES:
- See also: Related Info — http://www3.vghtc.gov.tw/tcm/english-index.htm